CLINICAL TRIAL: NCT03480633
Title: Preserved vs. Reduced Ejection Fraction Biomarker Registry and Precision Medicine Database for Ambulatory Heart Failure Patients (PREFER-HF) Study
Brief Title: Biomechanical Precision Medicine Registry for Patients With and Without Heart Failure
Acronym: PREFER-HF
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Hanna Kim Gaggin, Assistant Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2016P000339
Record Dates: First submitted 2018-02-22; First posted 2018-03-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure With Normal Ejection Fraction; Heart Failure With Reduced Ejection Fraction; Heart Failure, Right Sided; Heart Failure With Mid Range Ejection Fraction; Cardiovascular Risk Factor
Keywords: Heart failure; Precision medicine; High risk patients; Pathophysiology; Bioregistry; Biomarkers; Heart failure etiology
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Months
Biospecimen Retention: Samples With DNA — Blood samples will be collected at baseline as well as at 1 year follow up. At both time points, a total blood volume of up to 50 mL will be collected using EDTA and serum tubes, while patients are seated. Samples will be spun at 1800 rpm and plasma aliquoted. Samples will be frozen immediately at -80 C. For patients who opt to participate in the genetic portion of this study, buffy coat aliquoting and processing will be executed using the same blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Defined as patients without a history of heart failure
- Heart Failure w/NormalEjectionFraction: Heart Failure with Normal Ejection Fraction is defined as having a Left Ventricle Ejection Fraction of greater than or equal to 50%.
- HeartFailure w/ReducedEjectionFraction: Heart Failure with Reduced Ejection Fraction is defined as having a Left Ventricle Ejection Fraction of less than 50%.

SUMMARY:
In this single-center, longitudinal observational study, we will comprehensively examine clinical characteristics, proteomic, metabolomic, genomic and imaging data to better understand how different heart failure types may develop and progress over time. We will evaluate distinct sub-groups of heart failure (also known as heart failure phenotypes) and cardiomyopathies including amyloidosis with an ultimate goal of bringing the right medications and therapy to the right patients to optimize benefit and minimized side effects, an effort to improve precision medicine in heart failure.

DETAILED DESCRIPTION:
Patients 18-years and older with and without heart failure (across all left ventricular ejection fraction) and cardiomyopathies including amyloidosis will be enrolled in this single center, longitudinal observational Registry.

Baseline and one-year follow up blood samples including DNA as well as clinical characteristics, events leading up to heart failure diagnosis, etiology of heart failure, the presence and duration of other medical problems, laboratory, echocardiographic data and images, and therapy information will be obtained.

Clinical outcomes of interest include major adverse cardiovascular events (a combination of all-cause death and heart failure hospitalizations), individual endpoints of all-cause death, cardiovascular death, all-cause hospitalization, cardiovascular hospitalization, heart failure hospitalization, right-sided heart failure, and kidney injury.

Results from the Preserved vs. Reduced Ejection Fraction Biomarker Registry and Precision Medicine Database for Ambulatory Heart Failure Patients (PREFER-HF) trial will comprehensively examine longitudinal clinical characteristics, proteomic, metabolomic, genomic and imaging data to better understand pathophysiology of heart failure and phenotypes in heart failure with an ultimate goal of improving precision medicine in heart failure.

ELIGIBILITY:
Inclusion criteria for patients with HF:

* 18 years and older
* History of clinical symptoms consistent with HF and at least one of the following supporting evidence of HF:

  * NT-proBNP > 125 pg/mL
  * BNP > 35 pg/mL
  * Capillary wedge pressure ≥ 15 mmHg on right heart catheterization or CI <2.8 L/min/m2
  * LVEDP ≥ 15 mmHg
  * Radiographic evidence of pulmonary edema
  * Improvement in symptoms with diuretic initiation of increase
  * CPET evidence of cardiac etiology of symptoms

HFpEF: LVEF ≥ 50% HFrEF: LVEF <50%

Exclusion criteria (for all patients, including both those with HFpEF and HFrEF):

- End stage renal disease on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be identified and screened in inpatient units, via medical records, outpatient clinics, primary physician or specialist schedules, and through Research Patient Data Registry (RPDR).
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2016-04-07 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | Time from sample collection until the date of documented event up to 60 months after the study closure.
  MACE as defined by a combined end point of all-cause mortality and HF hospitalizations.

SECONDARY OUTCOMES:
Time to event: all-cause mortality | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.
Time to event: cardiovascular mortality | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.
Time to event: all-cause hospitalization | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.
Time to event: cardiovascular hospitalization | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.
Time to event: HF hospitalization | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.
Time to event: Right-sided HF | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.
Time to event: acute kidney injury | Time from sample collection until the date of documented event up to 60 months after the study closure.
  Medical records and phone follow-up with patients and/or their physicians will allow the investigators to ascertain vital status and any significant clinical events.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Gaggin, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abboud A, Nguonly A, Bean A, Brown KJ, Chen RF, Dudzinski D, Fiseha N, Joice M, Kimaiyo D, Martin M, Taylor C, Wei K, Welch M, Zlotoff DA, Januzzi JL, Gaggin HK. Rationale and design of the preserved versus reduced ejection fraction biomarker registry and precision medicine database for ambulatory patients with heart failure (PREFER-HF) study. Open Heart. 2021 Oct;8(2):e001704. doi: 10.1136/openhrt-2021-001704. PMID 34663746